CLINICAL TRIAL: NCT06770439
Title: A Phase II Study to Evaluate the Safety, Tolerability, and Efficacy of IBI343 Combined With Chemotherapy in Advanced Pancreatic Cancer
Brief Title: IBI343 Combined With Chemotherapy in Advanced Pancreatic Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, The president of the hospital, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CISPD-8
Record Dates: First submitted 2025-01-07; First posted 2025-01-13 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Advanced Pancreatic Cancers

STUDY DESIGN:
Intervention Model Description: There are two parts in this study, Part1 (safe lead-in phase) and Part2 (extension phase). In part1, patients with CLDN18.2-positive advanced pancreatic adenocarcinoma who had or had not previously received systemic therapy will be enrolled. The starting dose of the AG regimen was albumin-paclitaxel 100mg / m2 combined with gemcitabine 800mg / m2 by intravenous infusion (Intravenous, IV) D1 and D8 Q3W. If none of the first 3 subjects at 6 mg / kg had DLT during the DLT observation period, the combined high dose AG regimen was attempted. The investigator will adjust the dose of IBI343 combination chemotherapy according to the previous safety results and determine the safety of the combination dose, then entering the Part 2.
  In part2, 40 patients with CLDN18.2-positive advanced PDAC will be enrolled, 1:1 randomized to Arm A and Arm B, respectively. In Arm A, patients will receive IBI343 TBD + AG regimen (TBD); and in Arm B, patients will receive AG regimen.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental): In part1, patients with CLDN18.2-positive advanced pancreatic adenocarcinoma who had or had not previously received systemic therapy will be enrolled. The starting dose of the AG regimen was albumin-paclitaxel 100mg / m2 combined with gemcitabine 800mg / m2 by intravenous infusion (Intravenous, IV) D1 and D8 Q3W. If none of the first 3 subjects at 6 mg / kg had DLT during the DLT observation period, the combined high dose AG regimen was attempted. The investigator will adjust the dose of IBI343 combination chemotherapy according to the previous safety results and determine the safety of the combination dose, then entering the Part 2.
  Interventions: Drug: IBI343; Drug: Gemcitabine+Albumin-bound paclitaxel
- Part 2: Arm A (Experimental): In part2, 40 patients with CLDN18.2-positive advanced PDAC will be enrolled, 1:1 randomized to Arm A and Arm B, respectively. In Arm A, patients will receive IBI343 TBD + gemcitabine TBD + albumin-bound paclitaxel TBD.
  Interventions: Drug: IBI343; Drug: Gemcitabine+Albumin-bound paclitaxel
- Part 2: Arm B (Active Comparator): In part2, 40 patients with CLDN18.2-positive advanced PDAC will be enrolled, 1:1 randomized to Arm A and Arm B, respectively. In Arm B, patients will receive gemcitabine 1000mg / m2 d1, d8 Q3W + albumin-bound paclitaxel 125mg / m2d1, d8 Q3W treatment.
  Interventions: Drug: Gemcitabine+Albumin-bound paclitaxel

INTERVENTIONS:
Drug: IBI343 — IBI343 is a recombinant anti-tight junction protein 18.2 monoclonal antibody - ecotecan conjugate
  Arms: Part 1; Part 2: Arm A
Drug: Gemcitabine+Albumin-bound paclitaxel — Gemcitabine+ Albumin-bound paclitaxel is one of the recommended first line regime for advanced pancreatic cancer

SUMMARY:
This study is a phase II study to evaluate the safety, tolerability and efficacy of IBI343 combined with chemotherapy in patients with advanced pancreatic cancer, including Part1 (safe lead-in phase) and Part2 (extension phase). In part1, patients with CLDN18.2-positive advanced pancreatic adenocarcinoma who had or had not previously received systemic therapy were treated with chemotherapy in IBI343 with AG regimen (albumin paclitaxel with gemcitabine). In part2, 40 patients with CLDN18.2-positive advanced PDAC will be enrolled, 1:1 randomized to Arm A and Arm B, respectively. In Arm A, patients will receive IBI343 TBD + gemcitabine TBD + albumin-bound paclitaxel TBD; and in Arm B, patients will receive gemcitabine 1000mg / m2 d1, d8 Q3W + albumin-bound paclitaxel 125mg / m2d1, d8 Q3W treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent, willing and able to comply with the protocol specified visits and related procedures.
* Histopathologically confirmed unresectable locally advanced, recurrent, or metastatic pancreatic adenocarcinoma.
* Subjects must not be eligible for radical treatment such as radical radiotherapy and / or surgery; time to disease recurrence / metastasis> 6 months for subjects with previous (new) adjuvant / adjuvant / radiotherapy) chemotherapy / radical chemoradiotherapy. In part 1: locally advanced or recurrent / metastatic stage with or without systemic therapy (including chemotherapy, targeted therapy, tumor immunotherapy, etc.). In part 2: The locally advanced or recurrent / metastasis phase has not received any systemic therapy (including chemotherapy, targeted therapy, tumor immunotherapy, etc.).
* At least 1 measurable lesion (no previous radiotherapy) for solid tumors RECIST v1.1.(At baseline, computed tomography or magnetic resonance imaging showed the long diameter of 10 mm (except for lymph nodes, the short axis of the lymph node must be 15 mm), the diameter of the target lesion is 2 times the imaging layer thickness and the lesion is suitable for repeated accurate measurement. If a lesion located in the previously irradiated area clearly demonstrates a progression meeting the RECIST V1.1 criteria, the lesion acts as a measurable lesion).
* Age was 18 years, and gender was unlimited.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) was 0 or 1.
* The expected survival period was estimated at 12 weeks.
* Sufficient bone marrow and organ function.
* Female subjects of childbearing age or male partners of childbearing age should take effective contraception throughout the treatment period and within 6 months after the treatment period.
* Pathological tissue testing was confirmed as CLDN18.2 positive.

Exclusion Criteria:

* Is participating in another interventional clinical study, except for an observational (non-interventional) clinical study or is in the survival follow-up phase of the interventional study.
* Treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor within 2 weeks or 5 half-lives (whichever is longer) before the first dose of the study drug.
* The last anti-tumor therapy within 4 weeks before the first dose of the study drug or within 5 half-lives of the anti-tumor treatment (whichever is shorter) (2 weeks for washout with no exact half-life).
* Received therapeutic or palliative radiotherapy within 2 weeks prior to the first administration of the study drug.
* Receiving biliary stenting or PTCD within 7 days prior to the first use of study drug.
* Other anti-tumor treatment is planned during the study medication [allows palliative radiotherapy for the purpose of relieving symptoms (e. g. pain) and does not affect efficacy evaluation].
* Any live vaccine is administered within 4 weeks before the first dose of the study drug or during the duration of the study.
* A major surgical procedure (craniotomy, otomy, or tomy or otherwise defined by the investigator, excluding needle biopsy within 4 weeks before the first dose of study drug) or the presence of an unhealed wound, ulcer, or fracture; or a requirement that major surgery is planned during the study. For the purpose of palliative care, the local surgical treatment of isolated lesions is acceptable.

Any live vaccine within 4 weeks before the first dose of the study drug or during the duration of the study.

* A major surgical procedure (craniotomy, otomy, or tomy or otherwise defined by the investigator, excluding needle biopsy within 4 weeks before the first dose of study drug) or the presence of an unhealed wound, ulcer, or fracture; or a planned major surgery required during the study. For the purpose of palliative care, the local surgical treatment of isolated lesions is acceptable.
* Failure to recover to grade 0 or 1 prior to the first dose of study drug of NCI CTCAE v5.0 (excluding alopecia, fatigue, pigmentation, and other conditions with no safety risk as judged by the investigator).
* A history of gastrointestinal perforation and / or fistula within 6 months prior to the first dose of study drug was not resolved by surgery. presence of pyloric obstruction and / or persistent recurrent vomiting (3 times within 24 hours).
* After gastrointestinal or tracheal lumen stenting.
* Symptomatic CNS metastasis. For subjects with asymptomatic brain metastases (i. e., no glucocorticoid treatment, 1.5 cm treatment) or stable brain metastases after treatment, all the following criteria were required to participate in this study: no meson, pons, cerebellum, meninges, medullary or spinal cord metastasis; remained clinically stable for at least 4 weeks, confirmed clinical evidence of no new or expanded brain metastases, and stopped corticosteroid and anticonvulsant therapy for at least 2 weeks before the first dose of study drug. Note: The CNS is not used as a target lesion.
* Bone metastases at risk of paraplegia.
* Interstitial lung disease requiring steroid hormone therapy, or a history of - interstitial lung disease, non-infectious pneumonia, severely impaired or uncontrolled lung function, such as pulmonary fibrosis, severe radiation pneumonitis, acute lung injury, or is suspected during screening.
* There are diseases that fail to control History of the other primary malignancies.
* A known medical history of immunodeficiency.
* History of allogeneic organ transplantation and allogeneic HSCT.
* Previous treatment with antibody drug conjugates based on topoisomerase inhibitors.
* For medicated subjects, there was a previous history of allergy to the appropriate drug or preparation.
* For subjects receiving medication, there are contraindications to the drug.
* There was a history of prior drug-related non-morbidity.
* Female subjects in pregnancy or lactation.
* Other investigators are not eligible for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-04-18 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Up to 2 years
  The proportion of patients who had tumor evaluated as PR according to RECIST1.1 criteria during the whole study.
Adverse Event | Up to 2 years.
  Safety evaluation，such as hematotoxicity, hepatotoxicity, and renal function lab test, done continuously during treatment and the level of serum creatinine will be evaluated by using CTCAE 5.0 during study.

SECONDARY OUTCOMES:
Progression-free Survival | Up to 2 years.
  The time from enrolled to disease pregression or death from any cause during the whole study.
Duration of Response | Up to 2 years.
  The time from the first assessment of the tumor as CR or PR to the first assessment of PD or death from any cause during the whole study.
Disease Control Rate | Up to 2 years.
  The proportion of patients who had tumor evaluated as PR or SD according to RECIST1.1 criteria during the whole study.
Time to Response | Up to 2 years.
  The time from the first treatment to the first assessment of the tumor as CR or PR during the whole study.
Overall Survival | Up to 2 years.
  The time from enrolled to death from any cause during the whole study.

OTHER OUTCOMES:
CLDN18.2 expression levels in tumor tissues | Up to 2 years.
  To evaluate the correlation of CLDN18.2 expression levels in tumor tissues and the efficacy of IBI343 combination therapy

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - First Affiliated Hospital of Zhejiang University Schlool of Medicine, Hangzhou, Zhejiang
  - the First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No